CLINICAL TRIAL: NCT02527239
Title: Prevalence of Pompe's Disease Amongst Patients With Unexplained Respiratory Muscle Weakness or Respiratory Failure
Brief Title: Prevalence of Pompe's Disease in Respiratory Clinics
Acronym: PURF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015LF006B
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Pompe's Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prospective observational study — Prospective observational study collecting data during a clinic vist including measurement of respiratory muscle strength, respiratory failure, lung function, physical performance and blood testing for enzymes related to Pompe's disease and muscle function.

SUMMARY:
Pompe's disease is a very rare condition which causes weakness of the respiratory muscles and may therefore cause symptoms of breathlessness or even respiratory failure, requiring the use of a ventilator at night. Recently a treatment for this condition has become available as well as a simple diagnostic test. However, we believe it is possible that there are patients with this condition who are presently undiagnosed attending respiratory clinics.

We would like to complete an observational study of patients with respiratory muscle weakness of an unknown cause, who are attending respiratory clinics at two London centres, to determine whether patients attending these services have undiagnosed Pompe's disease.

DETAILED DESCRIPTION:
Participation in the study will involve taking measurements of respiratory muscle strength, lower limb strength and collecting blood samples to test for enzymes which relate to Pompe's disease. These measures will be completed during a routine clinic visit. Participation will also involve the study coordinator accessing medical notes to gain information about disease history.

The study aims to collect information about the number of patients attending respiratory clinics with undiagnosed Pompe's disease and the characteristics of these patients so that other specialist services could use these criteria to identify patients who may benefit from investigations and treatment. If any participants are diagnosed with Pompe's disease and could benefit from treatment medical staff would refer them for treatment at local UK centres.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to home mechanical ventilation or other respiratory clinics:

who are over 18 years old with unexplained respiratory muscle weakness with breathlessness and/or type II respiratory failure which may be treated by a ventilator which is: unexplained by a known pulmonary disease, radiological abnormality or distortion of body hiatus (e.g scoliosis or massive obesity defined as BMI > 50 kg/m2), associated with a restrictive ventilatory defect or associated with unexplained muscle weakness.

Exclusion Criteria:

respiratory muscle weakness confirmed to be due to another cause known to have Pompe's disease at time of referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged over 18 presenting to respiratory clinics with respiratory muscle weakness of an unknown cause.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The prevalence of undiagnosed adult onset Pompes disease. This will be assessed through dry blood spot testing measuring α-glucosidase (GAA) deficiency and the Activity Ratio +/Acarbose. | 12 months
  dry blood spot testing

SECONDARY OUTCOMES:
CK levels | 12 months
  blood tests
Respiratory muscle strength | 12 months
  Using sniff nasal inspiratory pressure, spirometry in lying and sitting, maximal inspiratory and expiratory mouth pressure
Respiratory failure | 12 months
  Blood gases
Muscle weakness | 12 months
  performance on the short physical performance battery
Disease history | 12 months
  review of notes to establish duration of symptoms, time interval between presentation and referral to secondary care and any signs of respiratory failure or respiratory muscle weakness at presentation.